CLINICAL TRIAL: NCT06223373
Title: Blood Flow Restriction Therapy Following Acute Shoulder Injury Patients: Assessment of Efficacy in Return to Activity
Brief Title: Blood Flow Restriction Therapy Following Acute Shoulder Injury Patients
Acronym: BFR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: unable to finish the study prior to graduation from residency
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00103746
Record Dates: First submitted 2024-01-16; First posted 2024-01-25 (Actual); Results first posted 2025-11-04 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2024-11

CONDITIONS: Shoulder Injury
Keywords: Upper extremity injuries; muscle atrophy; tendinopathy
MeSH Terms: conditions — Shoulder Injuries; Muscular Atrophy; Tendinopathy | interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Intervention Model Description: patients who will be recruited into randomized into 1 of 2 study arms: 1) those undergoing rehabilitation using Blood Flow Restriction (BFR) pressurized per standard protocols in addition to our institutional rehabilitation protocol or 2) those undergoing rehabilitation using "sham BFR" as well as our institutional rehabilitation protocol.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Blood Flow Restriction (BFR) (Experimental): Blood Flow Restriction (BFR) pressurized per standard protocols in addition to our institutional rehabilitation protocol
  Interventions: Device: Blood Flow Restriction
- "sham" Blood Flow Restriction (BFR) (Sham Comparator): rehabilitation using "sham BFR" as well as our institutional rehabilitation protocol
  Interventions: Device: "sham" Blood Flow Restriction

INTERVENTIONS:
Device: Blood Flow Restriction — In the BFR group, the tourniquet will be pressurized to 50% limb occlusion pressure (LOP), which is the pressure necessary for occluding 50% of arterial limb flow in the upper extremity.
  Other Names: BFR
  Arms: Blood Flow Restriction (BFR)
Device: "sham" Blood Flow Restriction — In the sham BFR group, the tourniquet will be pressurized to 0% occlusion pressure, while maintaining enough pressure to keep the tourniquet in place.
  Arms: "sham" Blood Flow Restriction (BFR)

SUMMARY:
Atrophy and weakness of the shoulder are a common problem following treatment of a number of shoulder and elbow pathologies. Even with relatively short periods of reduced activity, the magnitude of muscle loss can be quite substantial.

DETAILED DESCRIPTION:
Blood flow restriction (BFR) therapy is one such therapeutic tool that has received increasing attention, which involves application of a pressurized tourniquet to the injured limb during rehabilitation that limits atrophy when performing strength training with weight that otherwise would not produce enough of a contraction to prevent muscular atrophy. To date, several studies have been performed on BFR therapy, however, the effect of therapy on ligamentous and tendinous injury in the upper extremity remain unclear as most studies have focused on muscular strengthening in healthy individuals and on lower extremity injuries distal to the tourniquet.

ELIGIBILITY:
Inclusion Criteria:

* injured patient with clinical and magnetic resonance imaging (MRI) consistent with a formal diagnosis of non-operative rotator cuff and/or biceps tendinopathy
* no prior upper extremity ipsilateral procedures or history of deep vein thrombosis
* those willing to be part of the study

Exclusion Criteria:

* patients younger than 18 or older than 55 years of age
* a history of revision surgery or prior ipsilateral upper extremity surgery
* concomitant ligamentous, tendinous, or cartilage injury that would alter postoperative rehabilitation protocol
* inability to comply with the proposed follow-up clinic visits
* patients lacking decisional capacity

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2024-04-13 (Actual); Primary Completion 2024-10-18 (Actual); Study Completion 2024-10-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristen Nicholson, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Blood Flow Restriction (BFR) | "Sham" Blood Flow Restriction (BFR)
Started | 1 | 2
Completed | 0 | 0
Not Completed | 1 | 2
Not completed — Lost to Follow-up | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Blood Flow Restriction (BFR) | "Sham" Blood Flow Restriction (BFR) | Total
Number analyzed (Participants) | 1 | 2 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (0) | 41.5 (10.6) | 42.3 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 1 | 1 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Shoulder Muscle Strength Analysis: External Rotation (ER) Peak Torque Average (60 Degrees/Second)
Description: measuring shoulder strength in injured and non-injured arms for both study groups using a Biodex testing machine - Low Score indicates low torque/strength, high score indicates high torque/strength
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: ft-lb (pound foot)
Arm/Group | Blood Flow Restriction (BFR) | "Sham" Blood Flow Restriction (BFR)
Number analyzed (Participants) | 1 | 2
ft-lb (pound foot) | 28.6 (0) | 13.1 (8.3)

2. Primary Outcome: Shoulder Muscle Strength Analysis: External Rotation (ER) Peak Torque Average (60 Degrees/Second)
Description: as for outcome 1
Time Frame: Week 6
Population: Follow up measure was never performed or recorded for 1 sham patient due to loss of follow up.
Measure: Mean (Standard Deviation); unit: ft-lb (pound foot)
Arm/Group | Blood Flow Restriction (BFR) | "Sham" Blood Flow Restriction (BFR)
Number analyzed (Participants) | 1 | 1
ft-lb (pound foot) | 23.2 (0) | 19.2 (0)

3. Primary Outcome: Shoulder Muscle Strength Analysis: External Rotation (ER) Peak Torque Average (180 Degrees/Second)
Description: Low Score indicates low torque/strength, high score indicates high torque/strength
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: ft-lb (pound foot)
Arm/Group | Blood Flow Restriction (BFR) | "Sham" Blood Flow Restriction (BFR)
Number analyzed (Participants) | 1 | 2
ft-lb (pound foot) | 19.0 (0) | 11.1 (5.9)

4. Primary Outcome: Shoulder Muscle Strength Analysis: External Rotation (ER) Peak Torque Average (180 Degrees/Second)
Description: Low Score indicates low torque/strength, high score indicates high torque/strength
Time Frame: Week 6
Population: Follow up measure was never performed or recorded for 1 sham patient due to loss of follow up.
Measure: Mean (Standard Deviation); unit: ft-lb (pound foot)
Arm/Group | Blood Flow Restriction (BFR) | "Sham" Blood Flow Restriction (BFR)
Number analyzed (Participants) | 1 | 1
ft-lb (pound foot) | 16.6 (0) | 13.9 (0)

5. Primary Outcome: Shoulder Muscle Strength Analysis: External Rotation (ER) Peak Torque Average (300 Degrees/Second)
Description: Low Score indicates low torque/strength, high score indicates high torque/strength
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: ft-lb (pound foot)
Arm/Group | Blood Flow Restriction (BFR) | "Sham" Blood Flow Restriction (BFR)
Number analyzed (Participants) | 1 | 2
ft-lb (pound foot) | 14.4 (0) | 7.0 (0.28)

6. Primary Outcome: Shoulder Muscle Strength Analysis: External Rotation (ER) Peak Torque Average (300 Degrees/Second)
Description: Low Score indicates low torque/strength, high score indicates high torque/strength
Time Frame: Week 6
Population: Follow up measure was never performed or recorded for 1 sham patient due to loss of follow up.
Measure: Mean (Standard Deviation); unit: ft-lb (pound foot)
Arm/Group | Blood Flow Restriction (BFR) | "Sham" Blood Flow Restriction (BFR)
Number analyzed (Participants) | 1 | 1
ft-lb (pound foot) | 11.2 (0) | 13.6 (0)

7. Primary Outcome: Shoulder Muscle Strength Analysis: Internal Rotation (IR) Peak Torque Average (60 Degrees/Second)
Description: Low Score indicates low torque/strength, high score indicates high torque/strength
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: ft-lb (pound foot)
Arm/Group | Blood Flow Restriction (BFR) | "Sham" Blood Flow Restriction (BFR)
Number analyzed (Participants) | 1 | 2
ft-lb (pound foot) | 23.2 (0) | 11.0 (9.5)

8. Primary Outcome: Shoulder Muscle Strength Analysis: Internal Rotation (IR) Peak Torque Average (60 Degrees/Second)
Description: Low Score indicates low torque/strength, high score indicates high torque/strength
Time Frame: Week 6
Population: Follow up measure was never performed or recorded for 1 sham patient due to loss of follow up.
Measure: Mean (Standard Deviation); unit: ft-lb (pound foot)
Arm/Group | Blood Flow Restriction (BFR) | "Sham" Blood Flow Restriction (BFR)
Number analyzed (Participants) | 1 | 1
ft-lb (pound foot) | 27.2 (0) | 9.9 (0)

9. Primary Outcome: Shoulder Muscle Strength Analysis: Internal Rotation (IR) Peak Torque Average (180 Degrees/Second)
Description: Low Score indicates low torque/strength, high score indicates high torque/strength
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: ft-lb (pound foot)
Arm/Group | Blood Flow Restriction (BFR) | "Sham" Blood Flow Restriction (BFR)
Number analyzed (Participants) | 1 | 2
ft-lb (pound foot) | 23.5 (0) | 15.6 (7.8)

10. Primary Outcome: Shoulder Muscle Strength Analysis: Internal Rotation (IR) Peak Torque Average (180 Degrees/Second)
Description: Low Score indicates low torque/strength, high score indicates high torque/strength
Time Frame: Week 6
Population: Follow up measure was never performed or recorded for 1 sham patient due to loss of follow up.
Measure: Mean (Standard Deviation); unit: ft-lb (pound foot)
Arm/Group | Blood Flow Restriction (BFR) | "Sham" Blood Flow Restriction (BFR)
Number analyzed (Participants) | 1 | 1
ft-lb (pound foot) | 26.7 (0) | 7.6 (0)

11. Primary Outcome: Shoulder Muscle Strength Analysis: Internal Rotation (IR) Peak Torque Average (300 Degrees/Second)
Description: Low Score indicates low torque/strength, high score indicates high torque/strength
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: ft-lb (pound foot)
Arm/Group | Blood Flow Restriction (BFR) | "Sham" Blood Flow Restriction (BFR)
Number analyzed (Participants) | 1 | 2
ft-lb (pound foot) | 23.5 (0) | 14.5 (2.3)

12. Primary Outcome: Shoulder Muscle Strength Analysis: Internal Rotation (IR) Peak Torque Average (300 Degrees/Second)
Description: Low Score indicates low torque/strength, high score indicates high torque/strength
Time Frame: Week 6
Population: Follow up measure was never performed or recorded for 1 sham patient due to loss of follow up.
Measure: Mean (Standard Deviation); unit: ft-lb (pound foot)
Arm/Group | Blood Flow Restriction (BFR) | "Sham" Blood Flow Restriction (BFR)
Number analyzed (Participants) | 1 | 1
ft-lb (pound foot) | 26.6 (0) | 6.6 (0)

13. Primary Outcome: Rotator Cuff Muscle Cross Sectional Area (CSA) Measurement: Supraspinatus
Description: Ultrasound will be used to quantify the changes in rotator cuff muscle and distal biceps cross-sectional area before and after therapy. The same multifrequency linear probe (7.5-9.0 MHz, Elegra; Siemens Medical Solutions, Erlangen, Germany) will be used throughout the study.
Time Frame: Baseline
Measure: Median (Standard Deviation); unit: cm2
Arm/Group | Blood Flow Restriction (BFR) | "Sham" Blood Flow Restriction (BFR)
Number analyzed (Participants) | 1 | 2
cm2 | 10.04 (0) | 7.29 (1.23)

14. Primary Outcome: Rotator Cuff Muscle Cross Sectional Area (CSA) Measurement: Supraspinatus
Description: as for outcome 13
Time Frame: Week 3
Population: Patient elected to do PT at home and was lost to follow up
Measure: Mean (Standard Deviation); unit: cm2
Arm/Group | Blood Flow Restriction (BFR) | "Sham" Blood Flow Restriction (BFR)
Number analyzed (Participants) | 1 | 1
cm2 | 10.15 (0) | 6.33 (0)

15. Primary Outcome: Rotator Cuff Muscle Cross Sectional Area (CSA) Measurement: Supraspinatus
Description: as for outcome 13
Time Frame: Week 6
Population: Patient elected to do PT at home and was lost to follow up
Measure: Mean (Standard Deviation); unit: cm2
Arm/Group | Blood Flow Restriction (BFR) | "Sham" Blood Flow Restriction (BFR)
Number analyzed (Participants) | 1 | 1
cm2 | 10.34 (0) | 6.48 (0)

16. Primary Outcome: Rotator Cuff Muscle Cross Sectional Area (CSA) Measurement: Infraspinatus
Description: as for outcome 13
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: cm2
Arm/Group | Blood Flow Restriction (BFR) | "Sham" Blood Flow Restriction (BFR)
Number analyzed (Participants) | 1 | 2
cm2 | 11.84 (0) | 11.48 (0.24)

17. Primary Outcome: Rotator Cuff Muscle Cross Sectional Area (CSA) Measurement: Infraspinatus
Description: as for outcome 13
Time Frame: Week 3
Population: Patient elected to do PT at home and was lost to follow up
Measure: Mean (Standard Deviation); unit: cm2
Arm/Group | Blood Flow Restriction (BFR) | "Sham" Blood Flow Restriction (BFR)
Number analyzed (Participants) | 1 | 1
cm2 | 11.89 (0) | 11.24 (0)

18. Primary Outcome: Rotator Cuff Muscle Cross Sectional Area (CSA) Measurement: Infraspinatus
Description: as for outcome 13
Time Frame: Week 6
Population: Patient elected to do PT at home and was lost to follow up
Measure: Mean (Standard Deviation); unit: cm2
Arm/Group | Blood Flow Restriction (BFR) | "Sham" Blood Flow Restriction (BFR)
Number analyzed (Participants) | 1 | 1
cm2 | 12.33 (0) | 11.76 (0)

19. Primary Outcome: Visual Analog Scale (VAS) for PAIN - Baseline Scores
Description: Patients will receive questionnaires (VAS) at Baseline, Week 6, 6 and 12 months after completing rehabilitation - The VAS score can be interpreted into categories of pain or symptom intensity:
  0-4 mm: No pain. 5-44 mm: Mild pain. 45-74 mm: Moderate pain. 75-100 mm: Severe pain.
Time Frame: Baseline
Population: 1 patient did not have any data collected at this field
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Blood Flow Restriction (BFR) | "Sham" Blood Flow Restriction (BFR)
Number analyzed (Participants) | 1 | 1
score on a scale | 3 (0) | 5 (0)

20. Primary Outcome: Visual Analog Scale (VAS) for PAIN - Week 6 Scores
Description: as for outcome 19
Time Frame: Week 6
Population: Patient elected to do PT at home and was lost to follow up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Blood Flow Restriction (BFR) | "Sham" Blood Flow Restriction (BFR)
Number analyzed (Participants) | 1 | 1
score on a scale | 0 (0) | 4 (0)

21. Primary Outcome: Visual Analog Scale (VAS) for PAIN - Month 6 Scores
Description: as for outcome 19
Time Frame: Month 6
Population: 1 patient elected to do PT at home and 1 patient had surgery
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Blood Flow Restriction (BFR) | "Sham" Blood Flow Restriction (BFR)
Number analyzed (Participants) | 1 | 0
Score on a scale | 0 (0) |

22. Primary Outcome: Visual Analog Scale (VAS) for PAIN - Month 12 Scores
Description: as for outcome 19
Time Frame: Month 12
Population: All patients lost to follow up, value never collected
Arm/Group | Blood Flow Restriction (BFR) | "Sham" Blood Flow Restriction (BFR)
Number analyzed (Participants) | 0 | 0

23. Primary Outcome: American Shoulder and Elbow Surgeons Standardized Shoulder Assessment Form (ASES) Baseline Scores
Description: The American Shoulder and Elbow Surgeons (ASES) shoulder score is a patient-completed assessment for shoulder function and pain, ranging from 0 to 100, with higher scores indicating better function. Scoring involves a 50-point pain component derived from a visual analog scale (VAS), and a 50-point functional component from 10 activities of daily living questions, which are then weighted and added for the final score
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Blood Flow Restriction (BFR) | "Sham" Blood Flow Restriction (BFR)
Number analyzed (Participants) | 1 | 2
score on a scale | 73 (0) | 42.5 (6.6)

24. Primary Outcome: American Shoulder and Elbow Surgeons Standardized Shoulder Assessment Form (ASES) Week 6 Scores
Description: as for outcome 23
Time Frame: Week 6
Population: Patient elected to do PT at home and was lost to follow up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Blood Flow Restriction (BFR) | "Sham" Blood Flow Restriction (BFR)
Number analyzed (Participants) | 1 | 1
score on a scale | 95 (0) | 42 (0)

25. Primary Outcome: American Shoulder and Elbow Surgeons Standardized Shoulder Assessment Form (ASES) Month 6 Scores
Description: as for outcome 23
Time Frame: Month 6
Population: 2 Sham patients lost to follow up and measure was never reported or collected.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Blood Flow Restriction (BFR) | "Sham" Blood Flow Restriction (BFR)
Number analyzed (Participants) | 1 | 0
score on a scale | 100 (0) |

26. Primary Outcome: American Shoulder and Elbow Surgeons Standardized Shoulder Assessment Form (ASES) Month 12 Scores
Description: as for outcome 23
Time Frame: Month 12
Population: Patient lost to follow up, value never collected -Patient lost to follow up, value never collected
Arm/Group | Blood Flow Restriction (BFR) | "Sham" Blood Flow Restriction (BFR)
Number analyzed (Participants) | 0 | 0

27. Primary Outcome: Disabilities of the Arm, Shoulder, and Hand Scale (DASH) Baseline Scores
Description: The DASH score for patients ranges from 0 to 100, with 0 representing no disability and 100 indicating the greatest possible functional impairment of the upper extremity. Patients answer a 30-item questionnaire on a five-point scale (0-4 or 0-5 depending on the scale used), rating their ability to perform tasks and their symptoms. The sum of the raw scores is then transformed into the final 0-100 DASH score
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Blood Flow Restriction (BFR) | "Sham" Blood Flow Restriction (BFR)
Number analyzed (Participants) | 1 | 2
score on a scale | 35.5 (0) | 62.6 (27.4)

28. Primary Outcome: Disabilities of the Arm, Shoulder, and Hand Scale (DASH) Week 6 Scores
Description: as for outcome 27
Time Frame: Week 6
Population: Patient elected to do PT at home and was lost to follow up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Blood Flow Restriction (BFR) | "Sham" Blood Flow Restriction (BFR)
Number analyzed (Participants) | 1 | 1
score on a scale | 0 (0) | 68.4 (0)

29. Primary Outcome: Disabilities of the Arm, Shoulder, and Hand Scale (DASH) Month 6 Scores
Description: as for outcome 27
Time Frame: Month 6
Population: 2 Sham patients lost to follow up and measure was never reported or collected.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Blood Flow Restriction (BFR) | "Sham" Blood Flow Restriction (BFR)
Number analyzed (Participants) | 1 | 0
score on a scale | 0 (0) |

30. Primary Outcome: Disabilities of the Arm, Shoulder, and Hand Scale (DASH) Month 12 Scores
Description: as for outcome 27
Time Frame: Month 12
Population: Patient lost to follow up, value never collected - Patient lost to follow up, value never collected
Arm/Group | Blood Flow Restriction (BFR) | "Sham" Blood Flow Restriction (BFR)
Number analyzed (Participants) | 0 | 0

31. Primary Outcome: GH Levels - Baseline
Description: Patients will receive the blood draws in the physical therapy clinic - ELISA will be used to quantify plasma levels
Time Frame: Baseline
Population: The lab test required to run these data is a 96+ well plate that costs nearly $1000+. Our department could not financially justify buying this test to analyze 3 data points that would not provide reliable data for publication. Therefore, this test was never performed or analyzed.
Arm/Group | Blood Flow Restriction (BFR) | "Sham" Blood Flow Restriction (BFR)
Number analyzed (Participants) | 0 | 0

32. Primary Outcome: GH Levels - Week 3
Description: Patients will receive the blood draws in the physical therapy clinic - ELISA will be used to quantify plasma levels
Time Frame: Week 3
Population: as for outcome 31
Arm/Group | Blood Flow Restriction (BFR) | "Sham" Blood Flow Restriction (BFR)
Number analyzed (Participants) | 0 | 0

33. Primary Outcome: GH Levels - Week 6
Description: Patients will receive the blood draws in the physical therapy clinic - ELISA will be used to quantify plasma levels
Time Frame: Week 6
Population: as for outcome 31
Arm/Group | Blood Flow Restriction (BFR) | "Sham" Blood Flow Restriction (BFR)
Number analyzed (Participants) | 0 | 0

34. Primary Outcome: IGF-1 Levels - Baseline
Description: Patients will receive the blood draws in the physical therapy clinic - ELISA will be used to quantify plasma levels
Time Frame: Baseline
Population: as for outcome 31
Arm/Group | Blood Flow Restriction (BFR) | "Sham" Blood Flow Restriction (BFR)
Number analyzed (Participants) | 0 | 0

35. Primary Outcome: IGF-1 Levels - Week 3
Description: Patients will receive the blood draws in the physical therapy clinic - ELISA will be used to quantify plasma levels
Time Frame: Week 3
Population: as for outcome 31
Arm/Group | Blood Flow Restriction (BFR) | "Sham" Blood Flow Restriction (BFR)
Number analyzed (Participants) | 0 | 0

36. Primary Outcome: IGF-1 Levels - Week 6
Description: Patients will receive the blood draws in the physical therapy clinic - ELISA will be used to quantify plasma levels
Time Frame: Week 6
Population: as for outcome 31
Arm/Group | Blood Flow Restriction (BFR) | "Sham" Blood Flow Restriction (BFR)
Number analyzed (Participants) | 0 | 0

37. Primary Outcome: IL-6 Levels - Baseline
Description: Patients will receive the blood draws in the physical therapy clinic - ELISA will be used to quantify plasma levels
Time Frame: Baseline
Population: as for outcome 31
Arm/Group | Blood Flow Restriction (BFR) | "Sham" Blood Flow Restriction (BFR)
Number analyzed (Participants) | 0 | 0

38. Primary Outcome: IL-6 Levels - Week 3
Description: Patients will receive the blood draws in the physical therapy clinic - ELISA will be used to quantify plasma levels
Time Frame: Week 3
Population: as for outcome 31
Arm/Group | Blood Flow Restriction (BFR) | "Sham" Blood Flow Restriction (BFR)
Number analyzed (Participants) | 0 | 0

39. Primary Outcome: IL-6 Levels - Week 6
Description: Patients will receive the blood draws in the physical therapy clinic - ELISA will be used to quantify plasma levels
Time Frame: Week 6
Population: as for outcome 31
Arm/Group | Blood Flow Restriction (BFR) | "Sham" Blood Flow Restriction (BFR)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Month 6
Arm/Group | Blood Flow Restriction (BFR) | "Sham" Blood Flow Restriction (BFR)
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/2
Other Adverse Events (participants affected / at risk) | 0/1 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-04-19): https://cdn.clinicaltrials.gov/large-docs/73/NCT06223373/Prot_SAP_001.pdf
  • Informed Consent Form (2024-02-28): https://cdn.clinicaltrials.gov/large-docs/73/NCT06223373/ICF_000.pdf